CLINICAL TRIAL: NCT05698277
Title: Automated Fetal Cardiac Function Parameters in Congenital Heart Disease
Brief Title: Automated Fetal Cardiac Function in Babies Affected by Heart Diseases
Status: Recruiting | Type: Observational
Sponsor: Anna Erenbourg (Other)
Collaborators: Centre Hospitalier de Mayotte (Other); Vittore Buzzi Children's Hospital (Other); San Salvatore Hospital of L'Aquila (Other); Institute for Maternal and Child Health IRCCS Burlo Garofolo (Unknown); Sheba Medical Center (Other Government); Clinic of Fetal Echocardiography, Medical Centre UJASTEK (Unknown)
Responsible Party: Sponsor-Investigator, Anna Erenbourg, Consultant in Obstetrics and Gynaecology, The University of New South Wales
Organization: The University of New South Wales (Other)
Other Study IDs: 2022/ETH00943
Record Dates: First submitted 2022-12-18; First posted 2023-01-26 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Defect; Cardiac Function
Keywords: Congenital Heart Diseases; Fetal Cardiac Function
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Singleton pregnancies affected by congenital heart disease
  Interventions: Diagnostic Test: Automated fetal cardiac function evaluation
- Controls: Singleton healthy pregnancies
  Interventions: Diagnostic Test: Automated fetal cardiac function evaluation

INTERVENTIONS:
Diagnostic Test: Automated fetal cardiac function evaluation — Evaluation of ultrasound parameters by automated algorithms.
  Ultrasound assessed parameters are:
  1. Pulsed wave Doppler Modified Left and Right Myocardial performance indices
  2. Spatio-temporal image correlation Tricuspid, Mitral and Septal Annular Plane Systolic Excursion

SUMMARY:
The goal of this international multicentre prospective observational cohort study with a nested case-control study is to test some automated fetal heart functional parameters in healthy babies compared to those affected by a congenital heart condition.

The main questions it aims to answer are:

* If there is a significant difference between the two populations of infants
* Whether these parameters could significantly improve the predictive value of actual cardiovascular profile score to predict hydrops Participants will be offered two automated cardiac function assessments between 27+6 and 29+6 gestational weeks and between 34+6 and 36+6 weeks of gestation. Functional parameters will be compared between the two study groups and evaluated over time.

DETAILED DESCRIPTION:
Investigation Plan

Participating patients will be offered a fetal cardiac function echocardiography between 27+6 and 29+6 weeks of gestation and another between 34+6 and 36+6 weeks.

At the stage patients will come in to carry out fetal cardiac function echocardiography they will already know whether the baby is affected by congenital heart disease since malformation screening is carried out between 18 and 20 gestational weeks and will have already been undertaken. In the remote case of detecting an undiagnosed fetal malformation during one of the research scans, patients will be reassured, and appointments arranged at Maternal and Fetal medicine (MFM) clinic for further consultation along with notification of to their own treating doctor.

Every participant will be assigned a study number following recruiting order of participation. De-identification will be undertaken at image acquisition by the doctors prior to image review by the engineers. Researchers will access an online patients' form system, collect the assigned patients' number and add the necessary outcomes information. Ultrasound images will be saved locally in the ultrasound machine by the same assigned patient's study number and uploaded to a specific Microsoft (OneDrive) folder created in Sydney. This data will be stored for a minimum of 5 years after publication, then the data record will be securely destroyed in accordance with the University of New South Wales (UNSW) Records Disposal processes.

The research ultrasound scans will be performed by a trained sonographer using either a clinical ultrasound system or a research ultrasound system that is Therapeutic Goods Administration (TGA) approved for research imaging. The machine used clinically is made by one of the common commercial manufacturers (in this case General Electric E10) and is an identical model to that used in the Department of Maternal and Fetal Medicine. The machine used for research porpoises is called Vantage 256 and it is manufactured by a private company in the United States (Verasonics). It uses the same fundamental electronic circuitry and transducer design as conventional commercial machines, and in fact uses the same transducers as the commercial machines. However, the way that the ultrasound is delivered differs. Instead of transmitting beams as used in conventional ultrasound machines, Verasonics scans the area of interest by unfocused waves, allowing high quality images with a limited number of compounded plane-waves, and reduced acquisition time.

Women will be placed in a semi-recumbent position, as standard for pregnancy ultrasounds. After routine biometry, the research fetal cardiac function ultrasound will be carried out.

Each fetal cardiac function examination will include the following parameters:

1. Fetal biometric parameters (biparietal diameter, head circumference, abdominal circumference, femur diaphysis length)
2. Standard fetal Doppler parameters (umbilical artery, medial cerebral artery, ductus venosus)
3. Fetal cardiac heart rate
4. Presence of pericardial effusion or hydrops
5. Cardiac morphometry - all measurements carried out at the end of diastole, with the exception of atrial dimensions measured in systole (at their maximum extension)

   * Heart/thorax area measurement
   * 4 heart chambers measurements (apical/basal 4-chambers view in 2D)
   * Atrial and ventricular areas (apical/basal 4-chambers view in 2D)
   * Ventricular and atrial sphericity calculation
   * Inter-ventricular septum and myocardial walls thickness measurement (transversal 4-chambers view in 2D or M-mode)
6. Cardiac contractility

   * Spatio-temporal image correlation (STIC) M-Mode stroke volume, ejection fraction and shortening fraction
   * Automated STIC Mitral Annular Plane Systolic Excursion (MAPSE), Tricuspid Annular Plane Systolic Excursion (TAPSE), Septal Annular Plane Systolic Excursion (SAPSE)
   * Automated Pulsed Wave Doppler (PWD) Left and Right modified myocardial performance index (Mod-MPI)
7. Atrioventricular valves' function evaluation

   * Cine-loop evaluation of correct opening and closing
   * Anterograde Colour Doppler without regurgitation
   * Pulsed Doppler evaluation of flow velocity (monophasic or biphasic)
   * Left and right E/A ratio calculation
   * If any regurgitation: peak velocity and duration quantified
8. Aorta outflow evaluation

   * Aorta artery measurement (at the level of valvular ring in systole)
   * Aortic flow evaluation (Colour Doppler evaluation of systolic peak velocity)
9. Pulmonary outflow evaluation

   * Pulmonary artery measurement (at the level of valvular ring in systole)
   * Pulmonary flow evaluation (Colour Doppler evaluation of systolic peak velocity)
10. V-sign evaluation

    * Confirmation of anterograde flow in the entire length of the arteries
    * Pulsatility index of aortic isthmus and ductus arteriosus

All fetal morphometric and functional cardiac parameters will be normalised to Z-score by gestational age where possible. Fetal cardiac volumes and 2D images with inadequate quality due to fetal movements, presence of acoustic shadows of fetal ribs or spine, and maternal breathing will be excluded. If hydrops develops, cardiovascular profile score will be added to the routine cardiac function exploration.

The study population will be followed up until delivery and discharge of both mother and neonate. Patients' information will be collected anonymously. Each patient's history will be evaluated and information about previous pregnancies (maternal or fetal diseases during pregnancy) and outcomes (type of delivery, maternal and neonatal conditions at birth, long-term outcome of the pregnancy) will be collected. Furthermore, investigators plan to collect information about the current pregnancy (maternal and fetal observations during pregnancy) and outcomes (type of delivery, maternal and neonatal conditions at birth and up to hospital discharge of both).

Study Procedure Risks

There is no increased risk related to participating in this study. The study uses conventional ultrasound machinery as used in routine fetal evaluation, with no alteration in power output (as defined by Thermal Index or Mechanical Index). The Verasonics research ultrasound system is also comparable to conventional ultrasounds in terms of risks.

Approximately 20-30 minutes scan duration is anticipated for acquisition of the necessary research data which is in keeping with standard ultrasound examinations, and the As Low As Reasonably Achievable (ALARA) principle conventionally applied in fetal imaging.

Sample Size Calculation

The primary outcome of the study is the difference in the mean of automated fetal functional cardiac parameters between CHD cases and controls. This will be analysed using a two-sample t-test.

To estimate the sample size, the most commonly applied fetal functional parameter was used, specifically the left ventricle MPI (LV-MPI) as a proxy of all the automated fetal cardiac parameters.

Due to the rarity of congenital heart disease, the sample size calculation was performed based on recruiting two controls for each case. Pooled across cases with isolated pulmonary valve stenosis (n = 16) and controls (n = 48), a previous work observed a standard deviation of 0.098 in LV-MPI measurements. Using this observed pooled Standard Deviation (SD), a total sample of 381 pregnancies (127 CHD + 254 controls) with completed measurements is required to achieve at least 80% power to detect a difference of 0.03 in mean LV-MPI, with a two-sided type I error rate of 5%.

Investigators acknowledge that some pilot data may be required to evaluate the limited number of pathological cases and therefore some approximations are necessary e.g. for standard deviation within the population. For this reason, investigators have aimed to recruit a larger number of participants (approximately 30%), 165 CHD and 330 Controls, allowing also for some patient exclusions due to patient drop out, difficulties in scanning due to fetal movements etc, and incomplete data sets.

The aim would be to recruit sufficient cases to be able to estimate if there is significant difference in terms of fetal cardiac function parameters between affected and not affected fetuses to inform further research.

Data Analysis Plan

Raw (radio-frequency) ultrasound data generated using the Verasonics will allow the researchers to analyse the signal/image processing that takes place prior to display, enabling refinement of this imaging technique.

Image analysis will be carried out first manually through optical evaluation and then through the use of mathematical algorithms which will recognise and analyse only high-quality images. This could be a limitation because automatically only high-quality images will be included (which is not representative of real clinical work) but also guarantees that parameters are collected only from almost perfect research material (showing true differences if they exist).

Ultrasound images will be analysed and cardiac function parameters interpreted by South Eastern Sydney Local Health District (SESLHD)/UNSW researchers based at the Royal Hospital for Women (RHW), Randwick. Images will be analysed by a team of fetal medicine doctors at Royal Hospital for Women and UNSW engineers to assure that algorithms are correctly applied to calculate fetal cardiac function parameters.

Comparisons of interest between cases and controls in baseline characteristics will be performed using two-sample t-tests, Wilcoxon rank-sum tests or Pearson Chi-squared tests, as appropriate.

Secondary outcomes comparing cases and controls at a single time point will be analysed in a similar way to the primary outcome, subject to checks of assumptions. Analyses of changes in fetal function parameters over time (i.e. between the 27+6-29+6 and 34+6-36+6 week scans), and the comparison of these changes between cases and controls will employ generalised linear mixed models, as appropriate for the parameter.

Logistic regression will be used to estimate the association between fetal cardiac parameters and the incidence of hydrops. Receiver-operating-characteristics-curve analysis will be carried out to assess functional cardiac parameters compared to the routinely used cardiovascular profile score to predict cardiac failure in fetuses with congenital heart disease.

Statistical analysis will be performed using SPSS version 22.0 (SPSS Inc., Chicago, Illinois (IL), USA).

For those cases without complete data acquisition (i.e. intending but not undertaking a second scan), analysis will take place for only the isolated value and not for any temporal change. Their single gestational data set of ultrasound measurements will still be included in analysis but excluded from any analysis of sequential change.

Data Safety and Monitoring Board

To assure high quality data collection, images will be collected at each participating centre by experienced fetal medicine doctors who have practiced fetal medicine for over 10 years. Each image will be stored securely. Data will be anonymised and monitored by researchers at SESLHD/UNSW. Researchers at UNSW will also review and complete data collection in case of missing data.

Our team from RHW will supervise and guarantee the quality of the data. Each participating centre will have a site researcher, a fetal cardiologist who will discuss and sign consent form, collect ultrasound images and relevant patients' data. The data collected will be uploaded and securely stored onto the UNSW platform.

Once ethical approval for each overseas center will be granted, UNSW team will download data from all centers, merge the information in a unique database and analyze them with the help of a statistician. UNSW team will be responsible for images analysis and data analysis. All the participants will then collaborate in drafting manuscripts for publication.

Outcome data will be accessed only by authorised researchers using an encrypted code for data protection. Final drafts for publication will be reviewed by all the authors from each research site.

Dissemination of results and publication policy

Results of the study will be published in peer-reviewed scientific journals, presentations at conferences or other professional forums. In any publication, patient privacy will be protected and presented in a de-identified manner.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the CHD Group are as follows: singleton pregnancies; gestational age between 19+6 and 36+6 weeks gestation, determined by the last menstrual period and confirmed by first trimester ultrasound; isolated congenital cardiac anomaly diagnosed.
* Inclusion criteria for the Control Group are as follows: singleton pregnancies; gestational age between 19+6 and 27+6 weeks gestation, determined by the last menstrual period and confirmed by first trimester ultrasound; no congenital cardiac anomaly diagnosed

Exclusion Criteria common to the 2 groups (Cases and Controls):

* Fetuses whose mothers have comorbidities that have been proven to potentially affect cardiac function including:

  * intrahepatic cholestasis
  * pre-gestational and gestational diabetes
  * preeclampsia
  * growth restricted fetuses defined as estimated fetal weight or abdominal circumference <3rd percentile for GA
* Fetuses with other structural extracardiac anomalies at ultrasound examination
* Fetuses affected by any diagnosed genetic abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women will be recruited from each participating centre during their second or third trimester morphology scan.
  The Control Group will be mostly recruited at the time of the second trimester morphology scan; the CHD Group during a second/third trimester anomaly scan with collaboration and referral from the hospital fetal cardiologist.
  Healthy patients will be approached in the waiting room after their second trimester ultrasound scan, offered to participate and given a copy of a patient information sheet and consent form.
  CHD patients will be approached and offered to participate after consultation with perinatal cardiologists. A week after the first contact, we will phone patients to verify their intention to take part and to organize the fetal cardiac function follow up.
Sampling Method: Non-Probability Sample
Enrollment: 495 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Automated PWD-MPI comparing fetuses affected by congenital heart disease (CHD) to reference values across the fetal healthy population. | Measurements undertaken within the range 27+6 - 29+6 gestational weeks
  Measure the difference in the mean absolute numerical value for PWD-MPI (expressed to 2 decimal places) between fetuses with CHD overall compared to healthy fetuses and then by subgroups of different CHDs.
Automated STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion comparing fetuses affected by congenital heart disease to reference values across the fetal healthy population. | Measurements undertaken within the range 27+6 - 29+6 gestational weeks
  Difference in absolute values for each of STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion between fetuses with CHD overall compared to healthy fetuses and then by subgroups of different CHDs.
Automated PWD-MPI comparing fetuses affected by congenital heart disease (CHD) to reference values across the fetal healthy population. | Measurements undertaken within the range 34+6 - 36+6 gestational weeks
  Measure the difference in the mean absolute numerical value for PWD-MPI (expressed to 2 decimal places) between fetuses with CHD overall compared to healthy fetuses and then by subgroups of different CHDs.
Automated STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion comparing fetuses affected by congenital heart disease to reference values across the fetal healthy population. | Measurements undertaken within the range 34+6 - 36+6 gestational weeks
  Difference in absolute values for each of STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion between fetuses with CHD overall compared to healthy fetuses and then by subgroups of different CHDs.
Automated PWD-MPI comparing fetuses affected by congenital heart disease (CHD) to reference values across the fetal healthy population. | Measurements undertaken within the range 27+6 - 29+6 gestational weeks and within the range 34+6 - 36+6 gestational weeks
  Difference in variation of the mean absolute value for PWD-MPI over time between fetuses with CHD overall compared to healthy fetuses and then by subgroups of different CHDs.
Automated STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion comparing fetuses affected by congenital heart disease (CHD) to reference values across the fetal healthy population. | Measurements undertaken within the range 27+6 - 29+6 gestational weeks and within the range 34+6 - 36+6 gestational weeks
  Difference in variation of absolute values for each of STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion between fetuses with CHD overall compared to healthy fetuses and then by subgroups of different CHDs.

SECONDARY OUTCOMES:
Predictive value of Modified Cardiovascular Profile Score in hydrops (Adding Automated PWD-MPI to the classical cardiovascular profile score). | Measurements undertaken within the range 27+6 - 29+6 gestational weeks.
  Difference in predictive values between Modified and Classical Cardiovascular Profile Score. Minimum score value is 0, Maximum score value is 12. Higher score means a better outcome.
Predictive value of Modified Cardiovascular Profile Score in hydrops (Adding Automated PWD-MPI to the classical cardiovascular profile score). | Measurements undertaken within the range 34+6 - 36+6 gestational weeks.
  Difference in predictive values between Modified and Classical Cardiovascular Profile Score. Minimum score value is 0, Maximum score value is 12. Higher score means a better outcome.
Predictive value of Modified Cardiovascular Profile Score in hydrops (Adding Automated STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion to the classical cardiovascular profile score). | Measurements undertaken within the range 27+6 - 29+6 gestational weeks.
  Difference in predictive values between Modified and Classical Cardiovascular Profile Score. Minimum score value is 0, Maximum score value is 12. Higher score means a better outcome.
Predictive value of Modified Cardiovascular Profile Score in hydrops (Adding Automated STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion to the classical cardiovascular profile score). | Measurements undertaken within the range 34+6 - 36+6 gestational weeks.
  Difference in predictive values between Modified and Classical Cardiovascular Profile Score. Minimum score value is 0, Maximum score value is 12. Higher score means a better outcome.
Predictive value of Modified Cardiovascular Profile Score in hydrops (Adding Automated PW-MPI and STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion to the classical cardiovascular profile score). | Measurements undertaken within the range 27+6 - 29+6 gestational weeks.
  Difference in predictive values between Modified and Classical Cardiovascular Profile Score. Minimum score value is 0, Maximum score value is 14. Higher score means a better outcome.
Predictive value of Modified Cardiovascular Profile Score in hydrops (Adding Automated PW-MPI and STIC Tricuspid, Mitral and Septal Annular Plane Systolic Excursion to the classical cardiovascular profile score). | Measurements undertaken within the range 34+6 - 36+6 gestational weeks.
  Difference in predictive values between Modified and Classical Cardiovascular Profile Score. Minimum score value is 0, Maximum score value is 14. Higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Erenbourg, MD, Principal Investigator — The University of New South Wales; Alec W Welsh, MD PhD, Study Director — The University of New South Wales
Locations (7):
- Royal Hospital for Women, Sydney, New South Wales, Australia
- Sheba Medical Center, Tel Aviv, Israel
- Italy (3):
  - San Salvatore Hospital L'Aquila, L’Aquila
  - Vittore Buzzi Children's Hospital, Milan
  - Institute for Maternal and Child Health IRCCS Burlo Garofolo, Trieste
- Centre Hospitalier de Mayotte, Mamoudzou, Mayotte
- Medical Center Ujastek, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) that underlie results will be shared with other researchers in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available from 6 months after publication.
Access Criteria: Data will be accessible online on request by researchers. Requests will be reviewed and evaluated by the Principal Investigator. Data will be available for meta-analyses involving the collection, checking, and re-analysis of the original data for each participant in each study.

REFERENCES:
- [Background] Wu W, He J, Shao X. Incidence and mortality trend of congenital heart disease at the global, regional, and national level, 1990-2017. Medicine (Baltimore). 2020 Jun 5;99(23):e20593. doi: 10.1097/MD.0000000000020593. PMID 32502030
- [Background] Crispi F, Sepulveda-Martinez A, Crovetto F, Gomez O, Bijnens B, Gratacos E. Main Patterns of Fetal Cardiac Remodeling. Fetal Diagn Ther. 2020;47(5):337-344. doi: 10.1159/000506047. Epub 2020 Mar 26. PMID 32213773
- [Background] Walter C, Soveral I, Bartrons J, Escobar MC, Carretero JM, Quirado L, Gomez O, Sanchez-de-Toledo J. Comprehensive Functional Echocardiographic Assessment of Transposition of the Great Arteries: From Fetus to Newborn. Pediatr Cardiol. 2020 Apr;41(4):687-694. doi: 10.1007/s00246-019-02279-w. Epub 2020 Jan 10. PMID 31919591
- [Background] Guirado L, Crispi F, Masoller N, Bennasar M, Marimon E, Carretero J, Gratacos E, Martinez JM, Friedberg MK, Gomez O. Biventricular impact of mild to moderate fetal pulmonary valve stenosis. Ultrasound Obstet Gynecol. 2018 Mar;51(3):349-356. doi: 10.1002/uog.17456. PMID 28295792
- [Background] Inamura N, Taketazu M, Smallhorn JF, Hornberger LK. Left ventricular myocardial performance in the fetus with severe tricuspid valve disease and tricuspid insufficiency. Am J Perinatol. 2005 Feb;22(2):91-7. doi: 10.1055/s-2005-837739. PMID 15731988
- [Background] Lasa JJ, Tian ZY, Guo R, Rychik J. Perinatal course of Ebstein's anomaly and tricuspid valve dysplasia in the fetus. Prenat Diagn. 2012 Mar;32(3):245-51. doi: 10.1002/pd.2939. PMID 22430722
- [Background] Wohlmuth C, Wertaschnigg D, Wieser I, Arzt W, Tulzer G. Tissue Doppler imaging in fetuses with aortic stenosis and evolving hypoplastic left heart syndrome before and after fetal aortic valvuloplasty. Ultrasound Obstet Gynecol. 2016 May;47(5):608-15. doi: 10.1002/uog.14885. Epub 2016 Apr 17. PMID 25914144
- [Background] Chen J, Xie L, Dai L, Yu L, Liu L, Zhou Y, Wu G, Qin F, Liu H. Right Heart Function of Fetuses and Infants with Large Ventricular Septal Defect: A Longitudinal Case-Control Study. Pediatr Cardiol. 2016 Dec;37(8):1488-1497. doi: 10.1007/s00246-016-1462-z. Epub 2016 Aug 25. PMID 27562129
- [Background] Natarajan S, Szwast A, Tian Z, McCann M, Soffer D, Rychik J. Right ventricular mechanics in the fetus with hypoplastic left heart syndrome. J Am Soc Echocardiogr. 2013 May;26(5):515-20. doi: 10.1016/j.echo.2013.02.001. Epub 2013 Mar 6. PMID 23473605
- [Background] Nawaytou HM, Peyvandi S, Brook MM, Silverman N, Moon-Grady AJ. Right Ventricular Systolic-to-Diastolic Time Index: Hypoplastic Left Heart Fetuses Differ Significantly from Normal Fetuses. J Am Soc Echocardiogr. 2016 Feb;29(2):143-9. doi: 10.1016/j.echo.2015.08.014. Epub 2015 Sep 26. PMID 26394829
- [Background] Chen Y, Lv G, Li B, Wang Z. Cerebral vascular resistance and left ventricular myocardial performance in fetuses with Ebstein's anomaly. Am J Perinatol. 2009 Apr;26(4):253-8. doi: 10.1055/s-0028-1103152. Epub 2008 Nov 20. PMID 19023852
- [Background] Khandoker AH, Al-Angari HM, Marzbanrad F, Kimura Y. Investigating fetal myocardial function in heart anomalies by Doppler myocardial performance indices. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:2197-2200. doi: 10.1109/EMBC.2017.8037290. PMID 29060332
- [Background] Axt-Fliedner R, Graupner O, Kawecki A, Degenhardt J, Herrmann J, Tenzer A, Doelle A, Willruth A, Steinhard J, Gembruch U, Bahlmann F, Enzensberger C; Fetal Cardiac Imaging Research Group, Germany. Evaluation of right ventricular function in fetuses with hypoplastic left heart syndrome using tissue Doppler techniques. Ultrasound Obstet Gynecol. 2015 Jun;45(6):670-7. doi: 10.1002/uog.14736. Epub 2015 May 11. PMID 25418127
- [Background] Graupner O, Enzensberger C, Wieg L, Willruth A, Steinhard J, Gembruch U, Doelle A, Bahlmann F, Kawecki A, Degenhardt J, Wolter A, Herrmann J, Axt-Fliedner R; Fetal Cardiac Imaging Research Group Germany. Evaluation of right ventricular function in fetal hypoplastic left heart syndrome by color tissue Doppler imaging. Ultrasound Obstet Gynecol. 2016 Jun;47(6):732-8. doi: 10.1002/uog.14940. PMID 26138790
- [Background] Pedra SR, Hornberger LK, Leal SM, Taylor GP, Smallhorn JF. Cardiac function assessment in patients with family history of nonhypertrophic cardiomyopathy: a prenatal and postnatal study. Pediatr Cardiol. 2005 Sep-Oct;26(5):543-52. doi: 10.1007/s00246-004-0688-3. PMID 16132314
- [Background] Clur SB, Vink AS, Etheridge SP, Robles de Medina PG, Rydberg A, Ackerman MJ, Wilde AA, Blom NA, Benson DW, Herberg U, Donofrio MT, Cuneo BF. Left Ventricular Isovolumetric Relaxation Time Is Prolonged in Fetal Long-QT Syndrome. Circ Arrhythm Electrophysiol. 2018 Apr;11(4):e005797. doi: 10.1161/CIRCEP.117.005797. PMID 29654130
- [Background] Yozgat Y, Kilic A, Ozdemir R, Karadeniz C, Kucuk M, Karaarslan U, Mese T, Unal N. Modified myocardial performance index is not affected in fetuses with an isolated echogenic focus in the left ventricle. J Matern Fetal Neonatal Med. 2015 Feb;28(3):333-7. doi: 10.3109/14767058.2014.916679. Epub 2014 May 22. PMID 24749803
- [Background] Acharya G, Pavlovic M, Ewing L, Nollmann D, Leshko J, Huhta JC. Comparison between pulsed-wave Doppler- and tissue Doppler-derived Tei indices in fetuses with and without congenital heart disease. Ultrasound Obstet Gynecol. 2008 Apr;31(4):406-11. doi: 10.1002/uog.5292. PMID 18340627
- [Background] Patey O, Carvalho JS, Thilaganathan B. Urgent neonatal balloon atrial septostomy in simple transposition of the great arteries: predictive value of fetal cardiac parameters. Ultrasound Obstet Gynecol. 2021 May;57(5):756-768. doi: 10.1002/uog.22164. PMID 32730671
- [Background] Crispi F, Valenzuela-Alcaraz B, Cruz-Lemini M, Gratacos E. Ultrasound assessment of fetal cardiac function. Australas J Ultrasound Med. 2013 Nov;16(4):158-167. doi: 10.1002/j.2205-0140.2013.tb00242.x. Epub 2015 Dec 31. PMID 28191192
- [Background] Acharya G, Archer N, Huhta JC. Functional assessment of the evolution of congenital heart disease in utero. Curr Opin Pediatr. 2007 Oct;19(5):533-7. doi: 10.1097/MOP.0b013e3282efd2a2. PMID 17885470
- [Background] Maheshwari P, Henry A, Welsh AW. The Fetal Modified Myocardial Performance Index: Is Automation the Future? Biomed Res Int. 2015;2015:215910. doi: 10.1155/2015/215910. Epub 2015 Jun 22. PMID 26185751
- [Background] Herling L, Johnson J, Ferm-Widlund K, Zamprakou A, Westgren M, Acharya G. Automated quantitative evaluation of fetal atrioventricular annular plane systolic excursion. Ultrasound Obstet Gynecol. 2021 Dec;58(6):853-863. doi: 10.1002/uog.23703. PMID 34096674
- [Background] Garcia-Canadilla P, Sanchez-Martinez S, Crispi F, Bijnens B. Machine Learning in Fetal Cardiology: What to Expect. Fetal Diagn Ther. 2020;47(5):363-372. doi: 10.1159/000505021. Epub 2020 Jan 7. PMID 31910421
- [Background] Liu Y, Chen S, Zuhlke L, Black GC, Choy MK, Li N, Keavney BD. Global birth prevalence of congenital heart defects 1970-2017: updated systematic review and meta-analysis of 260 studies. Int J Epidemiol. 2019 Apr 1;48(2):455-463. doi: 10.1093/ije/dyz009. PMID 30783674
- [Background] Cohn JN, Ferrari R, Sharpe N. Cardiac remodeling--concepts and clinical implications: a consensus paper from an international forum on cardiac remodeling. Behalf of an International Forum on Cardiac Remodeling. J Am Coll Cardiol. 2000 Mar 1;35(3):569-82. doi: 10.1016/s0735-1097(99)00630-0. PMID 10716457
- [Background] Tan CMJ, Lewandowski AJ. The Transitional Heart: From Early Embryonic and Fetal Development to Neonatal Life. Fetal Diagn Ther. 2020;47(5):373-386. doi: 10.1159/000501906. Epub 2019 Sep 18. PMID 31533099
- [Background] Peixoto AB, Bravo-Valenzuela NJ, Rocha LA, Araujo Junior E. Spectral Doppler, tissue Doppler, and speckle-tracking echocardiography for the evaluation of fetal cardiac function: an update. Radiol Bras. 2021 Mar-Apr;54(2):99-106. doi: 10.1590/0100-3984.2020.0052. PMID 33854264
- [Background] Donofrio MT, Moon-Grady AJ, Hornberger LK, Copel JA, Sklansky MS, Abuhamad A, Cuneo BF, Huhta JC, Jonas RA, Krishnan A, Lacey S, Lee W, Michelfelder EC Sr, Rempel GR, Silverman NH, Spray TL, Strasburger JF, Tworetzky W, Rychik J; American Heart Association Adults With Congenital Heart Disease Joint Committee of the Council on Cardiovascular Disease in the Young and Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Council on Cardiovascular and Stroke Nursing. Diagnosis and treatment of fetal cardiac disease: a scientific statement from the American Heart Association. Circulation. 2014 May 27;129(21):2183-242. doi: 10.1161/01.cir.0000437597.44550.5d. Epub 2014 Apr 24. PMID 24763516
- [Background] Wieczorek A, Hernandez-Robles J, Ewing L, Leshko J, Luther S, Huhta J. Prediction of outcome of fetal congenital heart disease using a cardiovascular profile score. Ultrasound Obstet Gynecol. 2008 Mar;31(3):284-8. doi: 10.1002/uog.5177. PMID 18253925
- [Background] Huhta JC. Diagnosis and treatment of foetal heart failure: foetal echocardiography and foetal hydrops. Cardiol Young. 2015 Aug;25 Suppl 2:100-6. doi: 10.1017/S104795111500089X. PMID 26377716
- [Derived] Erenbourg A, Barber T, Cecotti V, Faiola S, Fantasia I, Stampaljia T, Avnet H, Radzyminska-Chrusciel B, Meriki N, Welsh A. Fetal cardiac function in pregnancy affected by congenital heart disease: protocol for a multicentre prospective cohort study. BMC Pregnancy Childbirth. 2025 Jan 30;25(1):99. doi: 10.1186/s12884-025-07145-7. PMID 39885422

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT05698277/Prot_SAP_000.pdf
  • Informed Consent Form: CHD PREGNANCY (Cases) (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT05698277/ICF_001.pdf
  • Informed Consent Form: NORMAL PREGNANCY (Controls) (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT05698277/ICF_002.pdf